CLINICAL TRIAL: NCT06688708
Title: 30-day and Lasting Impacts on Utilizing a Novel Vibrating Foot Orthosis for Tactile Stimulation in Diabetic Peripheral Neuropathy: a Double-blind, Randomized, Sham-controlled Trial
Brief Title: Long-term Effects of Using a Novel Orthotic Insole for Tactile Stimulation in Diabetic Peripheral Neuropathy and Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Natapatchakrid Thimabut, Principal Investigator, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWUEC-661032
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Peripheral Neuropathy Type 2
Keywords: Diabetic Peripheral Neuropathy; Noise; Orthosis; Stochastic Resonance; Tactile; Vibration

STUDY DESIGN:
Intervention Model Description: Intervention 1: Use vibrating foot orthosis with tactile stimulation Intervention 2: Use vibrating foot orthosis without tactile stimulation
Who Masked: Participant, Investigator
Masking Description: Allocation concealment Participants and Investigators were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use vibrating foot orthosis with tactile stimulation (Experimental): 32 participants were assigned to use a vibrating foot orthosis (VFO) with tactile stimulation (using the VFO combined with a random 0-100 Hz square wave pulse stimulus with pseudorandom white noise via a stochastic resonance approach) at home for 30 days. Participants had to conduct intervention for 60 minutes a day. 90% VPT of each participant was chosen as the subthreshold stimulation level for tactile stimulation. Posttests were given by three consecutive appointments on the 1st day, the 15th day, and the 30th day.
  Participants had to meet a prosthetist and orthotist (PO) at the experimental site on the three consecutive appointments for posttest evaluation.
  After completing this intervention, participants were followed up the VPT level by evaluation every 7 days.
  Interventions: Device: Using vibrating foot orthosis with tactile stimulation
- Use vibrating foot orthosis without tactile stimulation (Sham Comparator): 32 participants were assigned to use the VFO without tactile stimulation (using the VFO with only vibration 100 Hz frequency ) at home for 30 days. Participants were blinded. Even though there was no tactile stimulation, the device still performed vibration.
  Posttests were given by three consecutive appointments on the 1st day, the 15th day, and the 30th day.
  Participants had to meet a PO at the experimental site on the three consecutive appointments for posttest evaluation. Noted, there was no follow-up after completing this intervention.
  Interventions: Device: Using vibrating foot orthosis without tactile stimulation

INTERVENTIONS:
Device: Using vibrating foot orthosis with tactile stimulation — Stimulating tactile sensation by using vibrating foot orthosis in conjunction with a random 0-100 Hz square wave pulse stimulus and pseudorandom white noise via a stochastic resonance approach.
  Other Names: Using vibrating foot orthosis in conjunction with a random 0-100 Hz square wave pulse stimulus and pseudorandom white noise via a stochastic resonance approach
  Arms: Use vibrating foot orthosis with tactile stimulation
Device: Using vibrating foot orthosis without tactile stimulation — Stimulating tactile sensation by using vibrating foot orthosis with only vibration 100 Hz freqency.
  Other Names: Using vibrating foot orthosis with only vibration 100 Hz freqency
  Arms: Use vibrating foot orthosis without tactile stimulation

SUMMARY:
1. This study had the objectives to investigate the long-term and remaining effects of using a novel vibrating foot orthosis for tactile stimulation in diabetic peripheral neuropathy (DPN).
2. The hypothesis of this study was using the VFO in conjunction with a random square wave pulse stimulus and pseudorandom white noise via a stochastic resonance could effectively improve tactile sensitivity and reduce vibration perception threshold (VPT).
3. Participants were recruited from the HRH Princess Maha Chakri Sirindhorn Medical Centre (Srinakharinwirot University), Ongkharak, Nakhon Nayok, Thailand.
4. 64 type 2 diabetes mellitus people with mild-to-moderate peripheral neuropathy were recruited.
5. Approach to participant: use purposive sampling by direct contact the patients who match the inclusion criteria.
6. Informed Consent Process: the information sheet was provided to participants, and the researcher explained the objectives of the study, the duration of the research, the research method, the dangers or potential effects of the research, including the benefits that might arise from the research and other methods of treatment in details. The participants had enough time and opportunity to ask questions until they had a good understanding. The researchers willingly answered questions without hiding them, until they satisfied. Then, the participants had to willingly sign a consent form prior to participate in the research project with voluntary.
7. The study protocol was approved by the Human Research Ethics Committee of Srinakharinwirot University (SWUEC-661032).
8. A randomized sham-controlled trial was conducted in this study. The experiments in this study were performed in a parallel design with random allocation and a double-blind strategy (blinded participants and investigators).
9. Baseline characteristics were assessed including: muscle strength by manual muscle testing, grading by the Medical Research Council; sensation by the Semmes-Weinstein monofilament test (5.07 gauge, 10 g pressure size) with 10-site examination; peripheral neuropathy by the Michigan neuropathy screening instrument; vibratory perception by a tuning fork (a graduated Rydel-Seiffer version); body mass index; circulatory system examination by palpating dorsalis pedis and posterior tibial pulse; pathology of diabetic foot; VPT by the Vibratory Sensory Analyzer: VSA-3000 (Medoc Ltd., USA).
10. VPT values were determined as the outcome parameter.
11. Statistical methods:

    * Quantitative data will be presented with median (mean) and standard deviation (SD).
    * Qualitative data will be presented with numbers and percentages.
    * An independent t-test will be used to compare the independent outcomes.
    * A paired t-test will be used to compare the dependent outcomes.
    * A repeated-measures ANCOVA will be used for between group comparisons.
    * A repeated-measures ANOVA will be used for within-group comparison.
    * MANCOVA will be used for analyzing the covariates' effect on the relationship between the independent grouping variables and the continuous dependent variables.
    * Cohen's d will be used to determine the effect sizes.
12. Ethical Consideration (1) All participants were provided with detailed project information prior to participation in the research project.

(2) While conducting experiments, evaluating, collecting research results, a prosthetist and orthotist (PO) and a physician will be with the participants at all times to prevent possible accidents/adverse events.

(3) If there is any harm from the research, free medical treatment will be provided.

(4) During research participation, all participants have the rights to withdraw at any time without the need to give reasons.

(5) All information obtained from the research project will be kept as a secret, and will be disclosed to the public for academic benefits without the participants' name.

13. Expectable benefits and applications

1. Using the novel VFO may lead to efficient treatment for neurorehabilitation in DPN.
2. The investigators hope that this low-cost VFO can offer advantages such as affordability, widespread use, and home-based applications.
3. The benefits of using the novel VFO that can improve tactile sensation on the plantar surface of the foot in diabetic peripheral neuropathy.
4. Employing the novel VFO can reduce VPT.
5. Using the novel VFO can help prevent diabetic foot ulceration (DFU), lessen a risk of DFU recurrence, and avoid lower limb amputation.
6. Applying the novel VFO may help restore and prolong tactile sensation.
7. Using the novel VFO may aid in slowing DPN deterioration and decreasing peripheral nervous system impairment.
8. Utilizing the VFO may help improve quality of life for DPN people.

14. Compensations for participants

* Payment was provided for those participants who attend throughout the study.
* All participants received a custom-made foot orthosis after completing the study.

DETAILED DESCRIPTION:
According to diabetic peripheral neuropathy (DPN), the significant complications include diabetic foot ulceration (DFU), an increase in vibration perception threshold (VPT), a decrease in tactile sensitivity, and lower limb amputation. A vibrating insole is a novel gadget that can help reduce VPT and improve tactile sensibility.

This research project aimed to study the effectiveness of using a novel vibrating foot orthosis (VFO) combined with a random 0-100 Hz square wave pulse stimulus and pseudorandom white noise for stimulating tactile sensation in DPN. The remaining effects had also been observed after 30 days of intervention.

*Participation in this research is voluntary. The volunteers who participated in the study had 4 appointments. In the 1st appointment, the volunteers underwent clinical assessment, baseline assessment, vibration perception evaluation, and foot casting for fabricating a foot orthosis. Participants had been informed of all necessary details of the study and learned how to use the VFO safely and correctly. The participants had to use the VFO at home for 60 minutes a day over 30 days. In the 2nd to 4th appointments (the 1st, 15th, and 30th days) participants had to conduct the interventions and posttest assessment at the experimental site. A prosthetist and orthotist (PO) performed the experiment and outcome evaluation.

The VFO was comprised of two major components: a vibration generator and a custom-made foot orthosis (CFO). The vibration generator was composed of two signal generator circuits: a random 0-100 Hz square wave pulse stimulus generator circuit and a pseudorandom white noise (PRWN) generator circuit. A random square wave pulse stimulus (0-100 Hz) and PRWN were integrated by using a stochastic resonance (SR) approach to become an integrated stimulus. A vibratory actuator was implanted into the CFO and received the integrated stimulus. When the integrated stimulation signals were delivered to the implanted actuators, the VFO would perform vibration to stimulate across the entire soles of the feet.

In the experiments, participants were instructed to abstain from taking any medications that influence the nervous system's upkeep and any vitamins, including vitamin B3, B6, B complex, and no drinking alcohol for 48 hours prior to starting the experiments. Besides, participants have kept up with their regular regimen of other diabetes medications. Before beginning the experiment, participants needed to keep their blood sugar levels stable to avoid hypoglycemia.

Participants were randomized into two interventions by a computer-generated program. Intervention 1 was using the VFO combined with the integrated stimulus for tactile stimulation at subthreshold level (90% VPT). Intervention 2 was using the VFO with only 100 Hz frequency vibration.

The PO performed the experiments, pretest/baseline evaluation, and posttest assessment. The PO opened the close-sealed envelope to assign the interventions to participants. The PO and a rehabilitation doctor monitored all participants throughout the experiment and the 30-day intervention.

VPT values at the 1st metatarsophalangeal joint (MTP), 5th MTP, and calcaneal area were assessed as the outcomes. The posttests were evaluated on the 1st, 15th, and 30th days.

VPT assessment was performed by the VSA-3000. In VPT assessment, participants placed their feet on the VSA-3000 pedestal and laid the 1st MTP, 5th MTP, and calcaneus on the tip of the VSA-3000 stylus without pressing. The stylus would raise vibration from zero to a level perceived by participants. When participants detected the vibration, they immediately pressed the stop mouse to halt the vibrating stylus. Then a VPT value was obtained, and the assessment was repeated five times to determine an average VPT value.

During the interventions, participants were assigned to take a seat in a backrest chair, and the angle of their knees to the ground was perpendicular. Then, they put their bare feet on the VFO with fastening Velcro straps or sandal shoes. Interventions were performed with a 60-minute period. The PO and doctor would check participants' vibration perception. If they felt any vibration from the VFO, they were obliged to notify the PO or doctor immediately. The interventions would be stopped, and participants would be appointed to reassess their VPT levels, and the PO would set a new subthreshold stimulation level for them in a renewed trial.

Participants of Intervention 1 group would ask for voluntarily participating in the follow-up of the remaining effects after completing use of the VFO with integrated stimulus. Importantly, they also had been approved by their physicians before continuing into the follow-up. In the follow-up, participants had to continue to abstain from taking neurological drugs throughout the follow-up period. VPT assessment by the PO would performed every 7 days. The follow-up would end when VPT exceeded baseline.

Electrical safety testing and risk management for medical devices were performed in accordance with EN IEC 60601-1, ISO 14971, and the protocol for permission on medical devices in Thailand by the Medical Device Control Division of the Food and Drug Administration of Thailand to ensure that the VFO was safe for use in patients and clinical trials.

0.9 power, a 2-sided significance level of 0.05, 20% dropout were used to calculate the sample size. 64 participants were required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus and peripheral neuropathy diagnosis
* Absence of foot problems such as ulcers, calluses, skin problems, etc.
* No muscle weakness
* Stability in neurological and vital signs
* Adequate cognitive and language skills to follow instructions
* Ability to sense vibration
* Ability to sit for at least 60 minutes

Exclusion Criteria:

* Musculoskeletal problem that makes it difficult to use vibrating foot orthosis, such as severe pain or joint contracture in any foot joints
* Mental disorders
* Hypersensitivity to material substances in vibrating foot orthosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Vibration Perception Threshold (VPT) | Immediate assessment after finish intervention
  Vibration perception threshold (VPT) is the lowest vibrational intensity required to perceive a vibration stimulus, and VPT is known to be impaired at an early stage in various neuropathies. VPT is critical in detecting diabetic peripheral neuropathy early; as a result, VPT is relevant to the risk of diabetic foot ulceration (DFU). Thus, VPT is an effective predictor of the risk of DFU and it could be used to target DFU for early detection and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Natapatchakrid Thimabut, Ph.D., Principal Investigator — Srinakharinwirot University
Locations (1):
- Srinakharinwirot University, Ongkharak, Changwat Nakhon Nayok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing 1 year and after publication for a period of 2 years. Access to the IPD and documents will be open on the IPDShare website with registration. The information will be freely available and can be used for any purpose. There will not be any review process or no Data Use Agreement will be necessary.
Supporting Information: Study Protocol
Time Frame: IPD and documents will be available for sharing 1 year and after publication for a period of 2 years.